CLINICAL TRIAL: NCT06832605
Title: Effectiveness and Cost-utility of Mindfulness-based Cognitive Therapy (MBCT) to Prevent Depressive Relapse or Recurrence in Spanish Adults With Recurrent Depressive Disorder: a Controlled Trial.
Brief Title: Bounce-Back From Depression
Acronym: BECOME
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Sant Joan de Déu (Other)
Collaborators: Carlos III Health Institute (Other Government)
Responsible Party: Principal Investigator, Jesus Montero Marin, Senior Researcher Miguel Servet (CP21/00080), Fundació Sant Joan de Déu
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PI23/00021
Record Dates: First submitted 2025-01-09; First posted 2025-02-18 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Depression - Major Depressive Disorder
Keywords: Depression; MBCT; Relapse/recurrence prevention; Cost-utility; RCT
MeSH Terms: conditions — Depression; Recurrence | interventions — Mindfulness-Based Cognitive Therapy; Therapeutics

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment as Usual (TAU) (Active Comparator): TAU is administered in current daily practice and is defined as instructing participants to consult their family doctor or usual healthcare professional, as they normally would, if they experience symptomatic deterioration or difficulties during the study.
  Interventions: Other: Treatment as Usual (TAU)
- MBCT self-help (Experimental): The 'MBCT self-help' is based on the book 'The Mindfulness Way: An 8-week plan to free yourself from depression and emotional stress'. The book presents the 8-week MBCT course as a self-help booklet. Participants are asked to guide themselves using the self-help book. The book provides elaborate and practical mindfulness guidelines that can be exercised each week, as well as questions to help with reflection, ways to check progress and valuable feedback from others who have undertaken this MBCT programme.
  Interventions: Behavioral: MBCT self-help
- Group MBCT (Experimental): Group MBCT' will follow the treatment manual "Mindfulness-Based Cognitive Therapy for Depression". Group MBCT' is a systematic training in mindfulness meditation techniques to teach participants skills to prevent relapse/recurrence of depression. Treatment includes weekly 2-hour classes over an 8-week period with home exercises, a full day of practice (6 hours long, adapted for online delivery), and 4 booster sessions offered every 3 months from the start of the programme.
  Interventions: Behavioral: MBCT group

INTERVENTIONS:
Behavioral: MBCT group — MBCT is a systematic training in mindfulness meditation techniques to teach participants skills to prevent relapse/recurrence of depression. Treatment includes weekly 2-hour classes over an 8-week period with home exercises, a full day of practice (6 hours long, adapted for online delivery), and 4 booster sessions offered every 3 months from the start of the programme.
  Standard pharmacological treatment usually provided to patients suffering depression.
  Other Names: Mindfulness Based Cognitive Therapy; Treatment as Usual (TAU)
  Arms: Group MBCT
Behavioral: MBCT self-help — The 'MBCT self-help' is based on the book 'The Mindfulness Way: An 8-week plan to free yourself from depression and emotional stress'. The book presents the 8-week MBCT course as a self-help booklet. Participants are asked to guide themselves using the self-help book. The book provides elaborate and practical mindfulness guidelines that can be exercised each week, as well as questions to help with reflection, ways to check progress and valuable feedback from others who have undertaken this MBCT programme.
  Standard pharmacological treatment usually provided to patients suffering depression.
  Other Names: Mindfulness Based Cognitive Therapy; Treatment as Usual (TAU)
  Arms: MBCT self-help
Other: Treatment as Usual (TAU) — Standard pharmacological treatment usually provided to patients suffering depression.
  Arms: Treatment as Usual (TAU)

SUMMARY:
Objectives: To analyse the effectiveness of adding: (i) mindfulness-based cognitive therapy (MBCT) delivered through 8 videoconference group sessions (group MBCT), and (ii) MBCT delivered through a self-help manual and 3 low-intensity group support sessions (beginning, middle, and end of the program) via videoconference (supported MBCT self-help) to treatment as usual (TAU, normally maintenance antidepressant medication), for the treatment of patients with recurrent depression, compared with TAU alone. Furthermore, we will assess the cost-utility of group MBCT vs. supported MBCT self-help vs. TAU alone, identifying potential predictors and moderators of response, and exploring the mechanisms through which the interventions exert effects.

Study design: Multicentre randomised controlled trial, with pre-post, 6- and 12-months follow-ups. Centres: Parc Sanitari Sant Joan de Déu (St. Boi de Llobregat), Hospital Universitario Miguel Servet (Zaragoza), and Hospital del Mar (Barcelona).

Participants: Adult patients (n=300) with recurrent depression and high risk of relapse will be randomly assigned to group MBCT, supported MBCT self-help, or TAU.

Primary outcome: time from randomisation to depressive relapse/recurrence at 12-month follow-up (DSM-5). Secondaries: residual symptoms, well-being, quality of life, costs, and quality-adjusted life years. Process measures: rumination, mindfulness, decentering, affectivity, and self-compassion.

Main statistical analyses: Hazard ratios will be calculated using survival analysis. Secondary outcomes, predictors, and moderators will be tested using regression-based approaches. Incremental cost-utility ratios and mediation path-analyses will be estimated. Acceptability will be evaluated using qualitative methods.

DETAILED DESCRIPTION:
Depression is a prevalent mental health disorder, affecting around 10% of the Spanish population at least once in their lifetime. It is a recurrent condition with significant personal and societal costs. Despite available treatments, more than half of those affected experience multiple relapses, with higher risks after each episode. In Spain, antidepressants are commonly used for relapse prevention, but many patients prefer psychological treatments due to the side effects and low adherence associated with medication.

Mindfulness-Based Cognitive Therapy (MBCT) is a psychological intervention designed to prevent depressive relapse. It involves weekly two-hour sessions over two months. In other countries, particularly in the English-speaking world, MBCT has been shown to reduce relapse risk by 25%, making it a promising alternative or complement to long-term antidepressant use. MBCT helps patients recognize early signs of depression and manage negative thoughts, preventing the onset of new episodes. It has gained recognition in countries like the UK, where it is recommended for recurrent depression in public healthcare systems.

However, the effectiveness of MBCT for relapse prevention has not yet been fully evaluated in Spain through randomized clinical trials. This project aims to determine whether MBCT, added to usual treatment (TAU), is more effective than TAU alone in preventing depressive relapse or recurrence in Spanish adults with recurrent depression. The study will evaluate both in-person group MBCT sessions via videoconference and self-help formats, exploring their cost-utility, psychological mechanisms, and patient characteristics to identify those most likely to benefit from the therapy.

The Bounce-Back from Depression multicentre project will shed light on the application of MBCT in the Spanish context for the prevention of depressive relapse/recurrence. The use of different delivery formats will provide information about effectiveness, scalability, and cost-benefit.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18.
* Diagnosis of recurrent major depressive disorder, with ≥ 2 previous major depressive episodes (MDD), in partial remission.
* Internet access (via smartphone and computer).
* Understanding of written and read Spanish language.

Exclusion Criteria:

* Current severe MDD, current/past psychosis, bipolar disorder, history of schizophrenia, schizoaffective disorder, organic mental disorder, current severe substance abuse, organic brain damage, pervasive developmental delay, persistent antisocial behaviour, persistent self-injury requiring clinical treatment or therapy.
* No experience in the use of new technologies (computers/smartphones).
* Previously completed mindfulness training or extensive experience in meditation (i.e., i.e., no experience in the use of new technologies).
* Concurrent psychotherapy.
* No experience in the use of new technologies (computers/smart phones).
* Previously completed mindfulness training or extensive meditation experience (i.e. courses, retreats, or regular meditation).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Time from randomisation to relapse or recurrence of major depression at 12-month follow-up | Through study completion, an average of 1 year after randomization
  The primary outcome will be the time from randomisation to relapse or recurrence of major depression at 12-month follow-up, assessed in a time-to-event analysis, with patients followed at 3 different intervals during the study period (post-treatment, as well as 6-month and 12-month follow-up after randomisation). The presence of depression between assessments will be assessed retrospectively according to the Longitudinal Interval Follow-up Evaluation (LIFE), a form of the Structured Clinical Interview for DSM-5 (SCID) designed for longitudinal studies.

SECONDARY OUTCOMES:
Hamilton Depression Rating Scale (HDRS) | Through study completion, an average of 1 year after randomization
  Depressive symptoms
Beck Depression Inventory II (BDI-II) | Through study completion, an average of 1 year after randomization
  Severity of depression
Positive and Negative Affect Schedule (PANAS) | Through study completion, an average of 1 year after randomization
  Positive and Negative Affect
Short Warwick-Edinburgh Mental Well-Being Scale (SWEMWBS) | Through study completion, an average of 1 year after randomization
  Mental well-being
EuroQoL-5D (EQ-5D-5L) | Through study completion, an average of 1 year after randomization
  Health-related quality of life
Client Service Receipt Inventory (CSRI) | Through study completion, an average of 1 year after randomization
  Use of health and social services

OTHER OUTCOMES:
Sociodemographic-clinical data | Through study completion, an average of 1 year after randomization
  Socio-demographic data will include self-reported sex, date of birth (age), ethnicity, marital status, number of children, cohabitation, employment status and satisfaction, economic situation and relevant negative life events in the previous 6 months.
  Clinical data include history of mental illness, vulnerability factors (number of previous major depressive episodes, age at first onset of depression, presence of previous severe, prolonged or resistant episodes, childhood adversity (Childhood Trauma Questionnaire-Short Form [CTQ-SF]), number of hospital admissions, number of suicide attempts (if any), family history of mental illness and suicide, previous psychiatric and/or psychological treatments, life disorganisation (e.g., inability to work), type and dosage of medication at baseline (if prescribed), and psychological treatments received (during the last year), inability to work), type and dosage of medication at baseline (if prescribed), and psychological treatments received
Brooding subscale of Ruminative Responses Scale-Short Form (RRS) | Through study completion, an average of 1 year after randomization
  Rumination
Five Facet Mindfulness Questionnaire-Short Form (FFMQ-SF) | Through study completion, an average of 1 year after randomization
  Mindfulness skills
Decentering subscale of Experiences Questionnaire (EQ) | Through study completion, an average of 1 year after randomization
  Decentring
Sussex-Oxford Compassion Scale (SOCS-S) | Through study completion, an average of 1 year after randomization
  Self-compassion
Ecological Momentary Assessment (EMA) | Daily for 8 weeks
  The m-Path platform will be used and once a day during the 8 weeks of treatment we will assess mood states.
Mindfulness-Based Interventions-Participants; Assessment of Teaching (MBI:PAT) | Up to 8 weeks
  Participants´ perspective on the competence of MBCT education
Mindfulness-Based Interventions Teaching Assessment Criteria (MBI-TAC) | Up to 8 weeks
  Participants´ perspective on the competence of MBCT education

CONTACTS AND LOCATIONS:
Overall Officials: Jesus Montero, PhD, Principal Investigator — Fundació Sant Joan de Déu
Locations (3):
- Spain (3):
  - Parc Sanitari Sant Joan de Déu (PSSJD), Sant Boi de Llobregat, Barcelona
  - Parc de Salut Mar, Barcelona
  - Hospital Universitario Miguel Servet, Zaragoza